CLINICAL TRIAL: NCT04944862
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Single Dose Study to Assess the Safety, Pharmacokinetics, and Clinical Effect of CDX-0159 in Patients With Prurigo Nodularis
Brief Title: A Study of CDX-0159 in Patients With Prurigo Nodularis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDX0159-04
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Prurigo Nodularis
Keywords: CDX-0159; barzolvolimab
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CDX-0159 1.5mg/kg (Experimental): CDX-0159 1.5mg/kg administered once
  Interventions: Biological: CDX-0159
- CDX-0159 3mg/kg (Experimental): CDX-0159 3.0 mg/kg administered once
  Interventions: Biological: CDX-0159
- Placebo (Placebo Comparator): Normal saline administered once
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: CDX-0159 — administered intravenously
  Other Names: barzolvolimab
  Arms: CDX-0159 1.5mg/kg; CDX-0159 3mg/kg
Drug: Normal saline — administered intravenously
  Arms: Placebo

SUMMARY:
The purpose of the study is to explore the safety, clinical effect, pharmacodynamics, and pharmacokinetics of CDX-0159 (barzolvolimab) in patients with Prurigo Nodularis.

DETAILED DESCRIPTION:
The purpose of the study is to explore the safety, clinical effect, pharmacodynamics, and pharmacokinetics of CDX-0159 (barzolvolimab) in patients with Prurigo Nodularis.

There is a screening period of up to 2 weeks, an 8-week double-blind treatment period and a 16-week follow-up period after treatment. Patients will receive one dose of CDX-0159 (barzolvolimab) or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females, 18 - 75 years old.
2. Diagnosis of Prurigo Nodularis by a dermatologist at least 3 months prior to Screening with:

   1. At least 20 PN nodules with bilateral distribution on both arms and/or both legs and/or both sides of the trunk at screening.
   2. An Investigators Global Assessment (IGA) score for PN ≥ 3 at screening and Baseline (Day 1).
3. Severe itch, defined as the mean of the daily worst itch NRS (WI-NRS) score of ≥ 7 during the 7-day period immediately prior to initiation of study treatment.
4. Documented history of inadequate response to prescription topical medications or for whom topical medications are medically inadvisable.
5. Willing to apply a topical moisturizer (emollient) twice daily throughout the study.
6. Both males and females of child-bearing potential must agree to use highly effective contraceptives during the study and for 150 days afterwards after treatment.
7. Willing and able to complete a daily symptom electronic diary for the duration of the study and adhere to the study visit schedule.

Key Exclusion Criteria:

1. PN due to neuropathy, psychiatric disorders or medications.
2. Unilateral lesions of prurigo (eg, only one arm affected)
3. Active unstable pruritic skin conditions in addition to PN.
4. Women who are pregnant or nursing.
5. Known hepatitis B or hepatitis C infection or active COVID-19 infection
6. Vaccination with a live vaccine within 2 months prior to study drug administration (subjects must agree to avoid vaccination during the study and for four months thereafter). NOTE: Inactivated vaccines are allowed such as seasonal influenza for injection. COVID-19 vaccination is allowed.
7. History of anaphylaxis.

There are additional criteria that your study doctor will review with you to confirm you are eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by the incidence and severity of adverse events | From Day 1 (first dose) to Day 169 (last follow-up visit)
  Safety and tolerability of multiple dose levels of CDX-0159 as determined by drug related adverse events

SECONDARY OUTCOMES:
Pharmacokinetic evaluation | From Day 1 (before first dose) to Day 169 (last follow-up visit)
  CDX-0159 serum concentrations will be measured at specified visits
Clinical effect of CDX-0159 on pruritus | From Day 1 (first dose) to Day 57 (week 8)
  The mean percent change from baseline to Week 8 in the weekly average score of worst intensity itch per a numeric rating scale. The Worst Itch-Numerical Rating Scale (WI-NRS) ranges from 0 = "no itch" to 10 ="worst imaginable itch" for their worst intensity prurigo nodularis itch in the preceding 24-hr period.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - Desert Sky Dermatology, Tempe, Arizona
  - University of Miami, Dermatology Clinical Trials Unit, Miami, Florida
  - Revival Research Institute, LLC, Troy, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Markowitz Medical/Optiskin, New York, New York
  - Central Sooner Research, Norman, Oklahoma
  - Center for Clinical Studies, LTD.LLP, Houston, Texas
- Germany (7):
  - Charité Centrum für Innere Medizin und Dermatologie, Institute of Allergology (IFA), Berlin
  - Katholisches Klinikum Bochum gGmbH, Dermatologische Studienambulanz, Bochum
  - Universitatsklinikum Carl Gustav Carus Dresden, Klinik und Poliklinik fur Dermatologie, Dresden
  - Universitätsklinikum Frankfurt Klinik für Dermatologie, Venerologie und Allergologie Klinische Forschung, Frankfurt
  - Universitätsklinikum Erlangen Hautklinik, Mainz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz Hautklinik, Clinical Research Center, Mainz
  - Universitaetsklinikum Muenster (UKM) - Klinik für Hautkrankheiten, Münster
- Poland (3):
  - MT Medic Specjalistyczna Praktyka Lekarska, Krosno
  - IP Clinic Sp. z o.o., Lodz
  - Centrum Medyczne Ginemedica, Wroclaw